CLINICAL TRIAL: NCT03322072
Title: Calypso Guided High Precision Stereotactic Ablative Radiosurgery for Lung Tumors Using Real-Time Tumor Tracking & Respiratory Gating: A Seamless Phase I/II Prospective Clinical Trial
Brief Title: Calypso Guided High Precision Stereotactic Ablative Radiosurgery for Lung TUmours Using Real-Time Tumour Tracking & Respiratory Gating
Acronym: GPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CancerCare Manitoba (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Dr. Julian Kim, Assistant Professor, CancerCare Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRIC 2017-014
Record Dates: First submitted 2017-10-17; First posted 2017-10-26 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer Stage I; Lung Cancer Stage II; Lung Cancer, Nonsmall Cell; Lung Cancer Recurrent; Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single arm prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Real-Time Position Transponder Beacons (Experimental): Patients in this arm will each be receiving 3 implanted real-time position transponder beacons (Calypso beacons)
  Interventions: Device: Real-Time Position Transponder Beacons

INTERVENTIONS:
Device: Real-Time Position Transponder Beacons — The anchored lung tracking beacons are passive electromagnetic transponder beacons which are placed immediately adjacent to a lung tumor using a bronchoscope. Three beacons will be placed in the small airways of the lung adjacent to the target tumor (within 3 cm of the tumor). Each beacon measures 2 mm in diameter and 8 mm in length and consists of a miniature electrical circuit that is encapsulated in a biocompatible glass capsule. Each beacon has an affixed five-legged anchoring system which expands to 5mm diameter once deployed. The Calypso transponder beacon is placed endobronchially using the working channel of a bronchoscope. Navigational bronchoscopy can be used to pre-plan the optimal location for each beacon to be placed within the airways by using a pre-bronchoscopy CT scan.

SUMMARY:
This is a single arm seamless phase I/II prospective cohort study. Patients with early stage Non-Small Cell Lung Cancer (T1-T2N0M0) or those with a single pulmonary metastasis of a known malignancy (either following radical treatment or systemic therapy) will be offered participation in this study. Participants will have three tumor locator beacons placed with a flexible bronchoscope in the small bronchial airways in proximity (<3cm) from their lung tumors. These tumor locator beacons will provide real-time positional data and will allow for smaller treatment volumes of Stereotactic Ablative Radiosurgery (SABR) and also allow for a specialized form of treatment delivery known as respiratory gated SABR. This is expected to result in higher precision radiotheapy delivery with less radiotherapy dose to healthy tissues which are in close proximity to the lung tumours.

DETAILED DESCRIPTION:
This trial is a seamless phase I/II prospective, single arm, cohort study.

Phase I of the trial will consist of two patients and will serve to conduct quality assurance assessments and to familiarize thoracic surgeons, radiation oncologists, and medical physicists at CancerCare Manitoba and Health Sciences Center in the use and work flow of the Health Canada approved endobronchial implanted real-time tumor tracking transponder beacons. Patients in phase I will undergo standard stereotactic ablative radiotherapy (SABR) of a lung tumor with prior endobronchial transponder beacon placement. For phase I, the transponder beacons will be used for comparative localization analyses and SABR treatment setup procedures will be carried out independent of transponder beacon data, however, transponder data will be collected in order to conduct, post-treatment, in vivo quality assurance assessments of beacon performance characteristics. Otherwise, the SABR treatment for phase I will consist of the currently accepted standard internal target volume based and standard image guided SABR.

Phase II of this trial will consist of 26 patients who will undergo a specialized form of SABR radiotherapy specifically designed to take full advantage of the real-time tumor tracking ability of the transponder beacons. Specifically, SABR in phase II will consist of smaller radiotherapy treatment volumes employing respiratory gating and smaller planning target volume expansion margins given the superior tumor location telemetry afforded by the beacons. Comparative dosimetric analyses contrasting the traditional ITV/PTV style treatments to those with reduced ITV/PTV margins achieved via Calypso guided SABR will be performed. Patient self-reported quality of life and toxicity assessments will be collected with the goal of facilitating power and sample size calculations for the design of a larger phase III randomized controlled trial of Calypso guided SABR treatment in the future

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years of age who is surgically inoperable, or refusing surgical management.
2. Tumor criteria (a patient must satisfy one of "a", "b" below to be eligible):

   1. AJCC 7th edition clinical T1aN0M0, T1bN0M0, or T2aN0M0 (<4cm) Non-small cell lung cancer (adenocarcinoma, squamous cell carcinoma, or NSCLC Not Otherwise Specified) of the middle or lower lobes of the lung*;
   2. A single pulmonary metastasis (<4cm) of a known primary malignancy of any histology involving the middle or lower lobes of the lung* (either metastatic failure to a single pulmonary site after primary radical treatment, metastatic progression to a single lung metastasis following palliative chemotherapy, or a single pulmonary metastatic lesion of newly diagnosed stage IV malignancy).

      * upper lobe tumors are eligible for trial participation if the tumor has a demonstrated tumor motion of ≥1 cm in any axis (as assessed by fluoroscopy at the time of bronchoscopy).
3. Confirmation of malignancy (a patient must satisfy one of "a", "b" below to be eligible):

   1. Tumors accessible by bronchoscopy, image-guided percutaneous biopsy, or other invasive staging methods require biopsy confirmation of malignancy.
   2. If a tumor is not amenable to a diagnostic biopsy, evidence of growth of the target tumor on serial imaging scans is necessary prior to enrollment. An increase in SUV of the target tumor on serial PET scans is also acceptable.
4. ECOG performance status of 0 to 2.
5. Minimum life expectancy of 6 months.
6. Deemed fit to undergo bronchoscopy by their participating thoracic surgeon
7. Deemed fit to undergo SABR by their participating Radiation Oncologist.
8. Respiratory function (a patient must satisfy both "a" and "b" below):

   1. Minimum FEV1 of 0.8 liters
   2. Minimum DLCO of 35% predicted.
9. Able to provide written informed consent and understand verbal instructions necessary for radiotherapy treatments.

Exclusion Criteria:

1. Tumors located < 1cm from the chest wall based on CT imaging.
2. Tumors located ≤ 2 cm from the proximal bronchial tree (see figure 7)
3. Patients who require supplemental oxygen at rest.
4. Patients who are unable to lie flat or still for a minimum of 30 minutes.
5. ECOG performance status 3 or 4.
6. Evidence of uncontrolled extra-thoracic metastatic disease (based on imaging or clinical findings).
7. Proven or suspected intrathoracic lymph node involvement.
8. Prior SABR to the target tumor.
9. Prior history of idiopathic pulmonary fibrosis, interstitial lung disease, or active collagen vascular disease (systemic lupus erythematosus, Rheumatoid arthritis, or Scleroderma)
10. Pregnancy.
11. Active pulmonary infection
12. Known hypersensitivity to nickel titanium (Nitinol)
13. Known Bronchiectasis of the small airways nearest to the tumor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2025-01-14 (Estimated); Study Completion 2025-01-14 (Estimated)

PRIMARY OUTCOMES:
Mean within patient difference in PTV volumes | Assessed Immediately prior to RT start
  Mean within patient difference in PTV volumes of standard non-gated SABR treatment compared to PTV volumes of gated SABR using Calypso based PTV margins

SECONDARY OUTCOMES:
Patient self-reported quality of life | 1, 2, and 3 year
  EORTC QLQ - LC13 questionnaire
Acute and late toxicity assessment using the Common Terminology Criteria for Adverse Events (CTCAE version 4.0) | 1, 2, and 3 year
  Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
RT doses to Thoracic Organs at Risk | Assessed Immediately prior to RT start
  Mean within patient difference in radiotherapy doses to thoracic Organs at risk
Tumour Local Control | 1, 2, and 3 year
  Local Control (RECIST version 1.1 criteria)
Progression Free Survival | 1,2, and 3 year
  Progression Free Survival
Overall Survival | 1,2, and 3 year
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Health Sciences Center, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03322072/Prot_SAP_000.pdf